CLINICAL TRIAL: NCT00481494
Title: Personality Characteristics and Compliance With Antiglaucoma Medication
Acronym: GDC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Other Study IDs: 4-2007-0092
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-05

CONDITIONS: Glaucoma
Keywords: Glaucoma; Drug compliance; Personality
MeSH Terms: conditions — Glaucoma; Medication Adherence

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Personality traits may influence to the drug compliance in glaucoma patients.

DETAILED DESCRIPTION:
In chronic diseases, especially asymptomatic at early stage, drug compliance has been reported as an important factor to control them. And personality traits are associated with the drug compliance. However, there was few study to consider this relationship. We want to find the association the personality characteristics and drug compliance in glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic glaucoma
* Topical anti-glaucoma medications

Exclusion Criteria:

* Oral glaucoma medications

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-05; Study Completion 2007-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chan Yun Kim, MD, PhD, Study Chair — Department of Ophthalmology, Yonsei University College of Medicine
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea